CLINICAL TRIAL: NCT02003300
Title: The Modified Foldes-Biro Equation Used in Patients Under General Anaesthesia for the Measurement of Oxygen and Anaesthetic Agent Uptake
Brief Title: An Improved Method for the Measurement of Oxygen and Anaesthetic Agent Uptake in Patients Using the Foldes-Biro Equation
Status: Completed | Type: Observational
Sponsor: Bayside Health (Other Government)
Responsible Party: Sponsor
Other Study IDs: 177/03; GE/ASA Research Grant, 2004 (Other Grant/Funding Number: GE/ASA Research Grant, 2004)
Record Dates: First submitted 2013-12-03; First posted 2013-12-06 (Estimated); Last update posted 2013-12-06 (Estimated); Status verified 2004-12

CONDITIONS: E03.155.197; E03.155.253
Keywords: Oxygen uptake; Anesthetic gas uptake

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary aim is to confirm the efficacy of a new non-invasive method for measuring the oxygen uptake during general anesthesia of patients undergoing surgery under cardiopulmonary bypass. The method has already been successfully tested in the laboratory under controlled conditions. In the patient group chosen, oxygen uptake is simultaneously calculated, for comparison purposes, from monitoring measurements made routinely as part of normal patient care in these cases, using a pulmonary artery catheter - an invasive technique from which severe complications occasionally arise, including death.

A secondary aim is to elucidate the time course of uptake of the anaesthetic vapor, isoflurane, during this kind of surgery.

DETAILED DESCRIPTION:
In a series of 30 patients undergoing cardiopulmonary bypass, the change in nitrogen concentration between fresh gas entering the anesthetic breathing system and the exhaust gas leaving it in an otherwise closed system is used to determine total gas uptake by the principle of insoluble gas dilution. Oxygen and anaesthetic agent uptakes are then automatically determined by a computer directly linked to a rapid gas analyzer, every 15 seconds.

As a control, oxygen is calculated using the reverse Fick method. Measured arterial and mixed venous oxygen saturations were used to do this, and the cardiac output which was determined by thermodilution.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing non-emergency procedures using cardiopulmonary bypass in whom pulmonary artery catheterization was to be performed for routine monitoring purposes, including mixed venous oxygen determinations and thermodilution cardiac output determinations.

Exclusion Criteria:

* High risk patients (ASA 4+)
* Acute lung injury, sepsis
* Tricuspid regurgitation
* Patients under 18 years of age
* Patients unable to give informed consent

Ages: 18 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2005-04; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
oxygen uptake | During surgery

CONTACTS AND LOCATIONS:
Overall Officials: Brian J Lithgow, MESc BE BSc, Study Director — Monash University Department of Electrical Engineering; Gavin JB Robinson, MB BS FANZCA, Principal Investigator — The Alfred, Bayside Health; Philip J Peyton, MB BS FANZCA, Study Director — The Austin Hospital
Locations (1):
- The Alfred, Melbourne, Victoria, Australia

REFERENCES:
- [Background] Biro P. A formula to calculate oxygen uptake during low flow anesthesia based on FIO2 measurement. J Clin Monit Comput. 1998 Feb;14(2):141-4. doi: 10.1023/a:1007413018732. PMID 9669452